CLINICAL TRIAL: NCT05151432
Title: Combined Effect of Pulsed Electromagnetic Field and Pulsed Ultrasound Therapy in Treating Knee Osteoarthritis
Brief Title: Effect of Pulsed Electromagnetic Field and Pulsed Ultrasound in Treating Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Ahmed Fayez Zehiry, Principal investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Horus_MSc_2021
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Osteo Arthritis Knee; Ultrasound Therapy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pulsed US + Exercise Group (Experimental): Twenty subjects will receive PUT, plus an exercise program.
  Interventions: Device: Pulsed Ultrasound; Other: Traditional exercise program
- Pulsed Electromagnetic + Exercise Group (Experimental): Twenty subjects will receive PEMF, plus an exercise program.
  Interventions: Device: Pulsed Electromagnetic field; Other: Traditional exercise program
- Pulsed US + Pulsed Electromagnetic + Exercise Group (Experimental): Twenty subjects will receive PUT, PEMF, plus an exercise program.
  Interventions: Device: Pulsed Ultrasound; Device: Pulsed Electromagnetic field; Other: Traditional exercise program
- Sham + Exercise group (Experimental): Twenty subjects will receive sham PEMF and sham PUT plus exercises program.
  Interventions: Other: Traditional exercise program; Device: Sham Pulsed US & Electromagnetic field

INTERVENTIONS:
Device: Pulsed Ultrasound — Active US therapy will be administered using a device 4cm², 1- MHz US with a sound-head area of effective 4cm, radiating area of 3.5 to a beam non-uniformity ratio of cm². 5:1, and a therapeutic dose of approximately 112.5J/ That is, the pulsed US will be delivered for 9.5 minutes with a peak intensity of 1W/cm² at a 20% duty cycle, to achieve a spatial-temporal average intensity of 0.2W
  Arms: Pulsed US + Exercise Group; Pulsed US + Pulsed Electromagnetic + Exercise Group
Device: Pulsed Electromagnetic field — The patient's knee will be placed between 2 plates coil applicator generating a magnetic field intensity of 1.5 mT and a frequency of 75Hz.
  Arms: Pulsed Electromagnetic + Exercise Group; Pulsed US + Pulsed Electromagnetic + Exercise Group
Other: Traditional exercise program — Stretching exercises, Isometric quadriceps exercise, Straight leg raising (SLR) exercise, Isometric hip adduction exercise, Hip abductor strengthening, Hip extensor strengthening, Hip external rotator strengthening
Device: Sham Pulsed US & Electromagnetic field — The patients will receive Sham Pulsed US & Electromagnetic field.
  Arms: Sham + Exercise group

SUMMARY:
This study will be carried out to combine the effect of PEMF and PUT on pain, function, and ROM in patients with knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most frequent illnesses in the world, affecting the knee joint in particular. Osteoarthritis of the knee is the most common cause of physical limitations and a decline in quality of life. OA of the knee affects 250 million individuals worldwide (3.6 percent of the population). According to the World Health Organization's study on the global burden of illness, knee OA is expected to become the eighth-most

Ultrasound is one of the most often utilized and misunderstood treatment techniques. Ultrasound can help in the treatment or rehabilitation of musculoskeletal problems when utilized appropriately. When it is administered wrongly, however, the therapy provides little benefit at best, and at worst, the desired physiological effects are restricted or hindered.

Electrotherapy is frequently used for the treatment of different musculoskeletal disorders, The most common types of electrotherapy are ultrasound (US), iontophoresis, laser therapy, electromagnetic therapy, and transcutaneous electrical nerve stimulation (TENS). To our knowledge, no previous clinical trials have combined the effectiveness of PEMF and PUST in the treatment of knee OA. Therefore, this study will be conducted to combine the efficacy of PEMF and PUST in the treatment of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with moderate unilateral knee OA according to the American College of Rheumatology criteria

   * Morning stiffness
   * Crepitus on knee motion
   * Bony tenderness
   * No palpable warmth.
2. a population of individuals (45-55 years old).
3. patients are not obese their body mass index (BMI) will be> 30kg/ m2.
4. with a diagnosis grade 2 radiographic severity according to the Kellgren/Lawrence scale. grading scale The severity of the disease was radiologically evaluated by an orthopedic knee specialist.

Exclusion Criteria:

Patients with the following criteria will be excluded from participating in this study:

1. if they had received an intra-articular injection of hyaluronic acid or corticoids during the six months prior to the study.
2. if they had a clinical history of orthopedic knee surgery, a skin disorder.
3. cardiovascular diseases, such as acute myocardial infarction, during the previous month, or uncontrolled arterial hypertension, acute-phase respiratory conditions.
4. or if they had been receiving another kind of physiotherapeutic treatment.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-07 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | at baseline and after 4 weeks of intervention
  Assessing the change in pain intensity using visual analogue scale which consists of a 10-cm line anchored at each end. Score of 10 means (Worest possible pain) while score of 0 means (No pain).
Dynamic balance | at baseline and after 4 weeks of intervention
  Assessing the change in Dynamic balance using timed up and go test. It will be used to asses patients functional mobility. The patient will be asked to rise from a standard armchair, walk at a safe and comfortable pace to a mark 3 m away, then return to a sitting position in the chair, using gait aids and chair armrests to assist with sit to stand as needed.
Range of motion of knee | at baseline and after 4 weeks of intervention
  Assessing the change in knee rane of motion using electrogoniometer.

SECONDARY OUTCOMES:
Pain, Stiffness and function | at baseline and after 4 weeks of intervention
  Assessing the change in Pain, Stiffness and function using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). It consists of three subscales regarding pain, stiffness, and physical function with five, two, and 17 questions, respectively. Answers for these 24 questions are scored on five-point Likert scales (none = 0, slight = 1, moderate = 2, severe = 3, extreme = 4) with total scores ranging from 0 to 96. Higher scores indicate greater disease severity.
Walking ability | at baseline and after 4 weeks of intervention
  Assessing the change in Walking ability using the 10-meter walk test.which is reliable and valid test in patients with OA , measuring the required time for walking on a standard flat surface of 10 m.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Fayez, Demonstrator, Principal Investigator — Horus University in Egypt
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Horus University, Egypt, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided